CLINICAL TRIAL: NCT02749591
Title: Comparative Hybrid Effects of Combining Botulinum Toxin Type A With Robot-assisted Training v.s. With Mirror Therapy for Stroke Patients With Upper Extremity Spasticity: A Randomized Controlled Study
Brief Title: Comparative Hybrid Effects of Combining BoNT-A With Robot-assisted or Mirror Therapy for U/E Spasticity Stroke Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-9732A3
Record Dates: First submitted 2016-04-07; First posted 2016-04-25 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: stroke rehabilitation; spasticity; Botulinum toxin type A injection; robot-assisted therapy; mirror therapy; randomized controlled trial
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; Botulinum Toxins; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Robot-assisted therapy (RT) (Experimental): After injection with Botulinum Toxin Type A, a schedule of robot-assisted therapy appointments will be established. Each intervention includes 45 minutes of robotic training and 30 minutes of training in functional activities.
  Interventions: Drug: Botulinum Toxin Type A; Other: Robot-assisted therapy
- Mirror therapy (MT) (Experimental): After injection with Botulinum Toxin Type A, a schedule of mirror therapy appointments will be established.The MT group will receive a 45-minute MT per session followed by 30 minutes of task-oriented functional training.
  Interventions: Drug: Botulinum Toxin Type A; Other: Mirror therapy
- Control Intervention (CI) (Active Comparator): After injection with Botulinum Toxin Type A, a schedule of control intervention appointments will be established.The CI group will receive 75-minute rehabilitation program, focusing on upper extremity training and including neurodevelopmental techniques, trunk-arm control, weight bearing by the affected arm, fine motor tasks practice, functional task practice, and practice on compensatory strategies for daily activities.
  Interventions: Drug: Botulinum Toxin Type A; Other: Control intervention

INTERVENTIONS:
Drug: Botulinum Toxin Type A — To inject Botulinum toxin type A on the spasticity upper extremity for stroke patients.Doses and muscles selected for BoNT-A injection are individualized on the basis of a number of factors, including the spasticity patterns, severity of spasticity, and treatment goals
  Other Names: Botulinum Toxin
Other: Robot-assisted therapy — After injecting Botulinum toxin type A on the spasticity upper extremity, the RT group will receive a 45 minutes of robotic training and 30 minutes of training in functional training.
  Arms: Robot-assisted therapy (RT)
Other: Mirror therapy — After injecting Botulinum toxin type A on the spasticity upper extremity, the MT group will receive a 45-minute MT per session followed by 30 minutes of task-oriented functional training.
  Arms: Mirror therapy (MT)
Other: Control intervention — After injecting Botulinum toxin type A on the spasticity upper extremity, the CI group will receive 75-minute rehabilitation program, focusing on upper extremity training and including neurodevelopmental techniques, trunk-arm control, weight bearing by the affected arm, fine motor tasks practice, functional task practice, and practice on compensatory strategies for daily activities.
  Arms: Control Intervention (CI)

SUMMARY:
The aim of this study will be to determine and compare the immediate and longer-term effects of combination of BoNT-A injection and mirror therapy vs combination of BoNT-A injection and robot-assisted therapy.

DETAILED DESCRIPTION:
The purpose of this project is to examine and compare the immediate and long-term effects of combined Botulinum toxin type A injection with mirror therapy (MT) and with bilateral robot-assisted (RT) in patients with spastic hemiplegic stroke. Spasticity, a common impairment after stroke, has a profound impact on activity and participation for patients. BoNT-A injection combined with rehabilitation training is recommended to enhance functional recovery for stroke patients with spasticity. Although the positive combination effects of BoNT-A with stretch, RT, and constraint-induced movement therapy were reported, the quality of the evidence was weak due to methodology limitations. In addition, patients with spasticity usually have lower motor function and worse sensory deficits than patients without spasticity. Designing the post BoNT-A injection rehabilitation program should consider the above issues. RT and MT are two interventions providing sensorimotor input for patient with low level of motor function. It is unknown whether combining BoNT-A injection with RT or with MT have positive effects and engenders differential effects on motor and related functional performance.

At least 60 participants with chronic spastic hemiplegic stroke will be recruited and randomly assigned to one of 3 groups: BoNT-A injection with RT, BoNT-A injection with MT, and BoNT-A injection with control intervention (CI). All the post-injection interventions will be implemented 60 minutes/day, 3 days/week, for 8 weeks. The RT group will receive 30-minute RT, followed by 30-minute functional training. The MT group will receive 30-minute MT, followed by 30-minute functional training. The CI group will receive 60-minute rehabilitation program, such as bilateral arm training and functional task practice. Body function and structures outcome measures include Fugl-Meyer Assessment, Modified Ashworth Scale, Medical Research Council scale, myometer (Myoton-3), actigraph, and Pittsburgh Sleep Quality Index. Activity and participation measures include Wolf Motor Function Test, Ten meter walk test, Motor Activity Log, Nottingham Extended Activities of Daily Living Scale, and Canadian Occupational Performance Measure. In addition, to directly reflect a patient's unique needs and goals, Goal Attainment Scaling will be assessed. Evaluators will be blind to group allocation. The outcome will be measured at pre-treatment, post-treatment, and 3-month follow-up.

This comparative efficacy study will be the first to examine and compare the immediate and long-term combination effects of BoNT injection with RT, MT, or CI. The follow-up assessments will provide the long-term effects of different treatments on health-related outcomes, which are crucial for community reentry. In addition, the results of objective assessments and patient-reported outcomes may lead to individualized upper limb training following BoNT-A injection for patients with spastic hemiplegic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Clinical and imagine diagnosis of a first or recurrent unilateral stroke ≥ 3 months
* Upper limb spasticity (Modified Ashworth scale of ≥ 2)
* Moderate to severe movement impairment of U/E (FMA score ranging from 18 to 56)
* No serious cognitive impairment (i.e., Mini Mental State Exam score > 18)
* Age ≥ 18 years

Exclusion Criteria:

* Pregnant
* Bilateral hemispheric or cerebellar lesions
* Significant visual field deficits or hemineglect
* Contraindication for BoNT-A injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Motor function assessed on Fugl-Meyer Assessment (FMA) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.

SECONDARY OUTCOMES:
Muscle power assessed on Medical Research Council Scale (MRC) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
Muscle tone assessed on Modified Ashworth Scale (MAS) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The functional state assessed on Myometer Assessment | Change from baseline at 5 months
  The outcome will be measured at 4 time points: 0 week, 1 week, 8 weeks, and 5 months after recruitment.
The amount of movement assessed on Actigraph Assessment | Change from baseline at 2 months
  The outcome will be measured at 2 time points: 0 week, and 8 weeks after recruitment.
The quality of sleep assessed on Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
Walking speed assessed on Ten Meter Walk Test (10MWT) | Change from baseline at 2 months
  The outcome will be measured at 2 time points: 0 week, and 8 weeks after recruitment.
The upper extremity motor ability assessed on Wolf Motor Function Test (WMFT) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The quality of movement and amount of use assessed on Motor Activity Log (MAL) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The instrumental activities of daily living assessed on Nottingham Extended Activities of Daily Living Scale (NEADL) | Change from baseline at 5 months
  The outcome will be measured at 3 time points: 0 week, 8 weeks, and 5 months after recruitment.
The participant's perception of the performance assessed on Canadian Occupational Performance Measure (COPM) | Change from baseline at 2 months
  The outcome will be measured at 3 time points: 0 week, 1week, and 8 weeks after recruitment.
The participants' individual goals assessed on Goal attainment scale (GAS) | Change from baseline at 5 months
  The outcome will be measured at 4 time points: 0 week, 1 week, 8 weeks, and 5 months after recruitment.
Revised Notttingham Sensory Assessment (RNSA) | Change from baseline at 2 months
  The outcome will be measured at 3 time points: 0 week, 1week, and 8 weeks after recruitment.
Stroke Impact Scale (SIS) | Change from baseline at 5 months
  The outcome will be measured at 4 time points: 0 week, 1 week, 8 weeks, and 5 months after recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Wen Hung, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Rehabilitation, Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ada L, O'Dwyer N, O'Neill E. Relation between spasticity, weakness and contracture of the elbow flexors and upper limb activity after stroke: an observational study. Disabil Rehabil. 2006 Jul 15-30;28(13-14):891-7. doi: 10.1080/09638280500535165. PMID 16777777
- [Result] Amano S, Takebayashi T, Hanada K, Umeji A, Marumoto K, Furukawa K, Domen K. Constraint-Induced Movement Therapy After Injection of Botulinum Toxin Type A for a Patient With Chronic Stroke: One-Year Follow-up Case Report. Phys Ther. 2015 Jul;95(7):1039-45. doi: 10.2522/ptj.20140329. Epub 2015 Jan 15. PMID 25592185
- [Result] Bhakta BB, Cozens JA, Chamberlain MA, Bamford JM. Impact of botulinum toxin type A on disability and carer burden due to arm spasticity after stroke: a randomised double blind placebo controlled trial. J Neurol Neurosurg Psychiatry. 2000 Aug;69(2):217-21. doi: 10.1136/jnnp.69.2.217. PMID 10896696
- [Result] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245